CLINICAL TRIAL: NCT04219358
Title: Evaluation of Topical Application of 5% Imiquimod, 0.05% Imiquimod and 0.05% Nanoencapsulated Imiquimod Gel in the Treatment of Actinic Cheilitis: a Randomized Controlled Trial
Brief Title: Topical Application of Imiquimod Gel at Different Concentrations in Actinic Cheilitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated because of COVID19 pandemics.
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-0656
Record Dates: First submitted 2019-10-04; First posted 2020-01-07 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Actinic Cheilitis
Keywords: imiquimod; nanoencapsulation
MeSH Terms: conditions — Actinic cheilitis | interventions — Imiquimod; Gels; dexpanthenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A pharmacist, who will not have contact with the study subjects at any time, will prepare the hydrogels in transparent sealed syringes, which will be numerically coded and two spreadsheets with the codes will be generated and placed in sealed brown envelopes. One envelope will be held by the pharmacist and the other envelope will be placed in a safe place. Participants will not know which medication they received until the end of the experimental phase. The vehicle gel is identical in appearance to those containing imiquimod. If for any reason the information on which treatment has been allocated is required, the external assistant will take all possible measures to ensure that the masking is not broken. The examiners who will perform the treatment and clinical evaluation will be blinded to the experimental group. Primary outcome measure is based on clinical evaluation of lesions by photographs. The images will be coded in order to achieve blindness of outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo & Standard Treatment (Active Comparator)
  Interventions: Drug: Vehicle Gel Base; Drug: Lip sunscreen 30 Sun Protector Factor (SPF); Drug: Dexpanthenol
- Imiquimod 5% & Standard Treatment (Experimental)
  Interventions: Drug: Imiquimod 5% gel; Drug: Lip sunscreen 30 Sun Protector Factor (SPF); Drug: Dexpanthenol
- Imiquimod 0.05% & Standard Treatment (Experimental)
  Interventions: Drug: Imiquimod 0,05% gel; Drug: Lip sunscreen 30 Sun Protector Factor (SPF); Drug: Dexpanthenol
- Imiquimod nanoencapsulated 0.05% & Standard Treatment (Experimental)
  Interventions: Drug: Imiquimod nanoencapsulated 0,05% gel; Drug: Lip sunscreen 30 Sun Protector Factor (SPF); Drug: Dexpanthenol

INTERVENTIONS:
Drug: Vehicle Gel Base — Apply 0.5ml of gel stored in a 1ml syringe over the lip 3 times a week (Mondays, Wednesdays and Fridays) at night for a period of 4 weeks.
  Gel components: medium molecular weight chitosan, lactic acid 85% and water.
  Arms: Placebo & Standard Treatment
Drug: Imiquimod 5% gel — Apply 0.5ml of gel stored in a 1ml syringe over the lip 3 times a week (Mondays, Wednesdays and Fridays) at night for a period of 4 weeks.
  Gel components: medium molecular weight chitosan, lactic acid 85% and free form imiquimod 5%.
  Arms: Imiquimod 5% & Standard Treatment
Drug: Imiquimod 0,05% gel — Apply 0.5ml of gel stored in a 1ml syringe over the lip 3 times a week (Mondays, Wednesdays and Fridays) at night for a period of 4 weeks.
  Gel components: medium molecular weight chitosan, lactic acid 85% and imiquimod 0.05% free form.
  Arms: Imiquimod 0.05% & Standard Treatment
Drug: Imiquimod nanoencapsulated 0,05% gel — Apply 0.5ml of gel stored in a 1ml syringe over the lip 3 times a week (Mondays, Wednesdays and Fridays) at night for a period of 4 weeks.
  Gel components: medium molecular weight chitosan, lactic acid 85% and imiquomod in a nanoencapsulated suspension at concentration of 0,05%
  Arms: Imiquimod nanoencapsulated 0.05% & Standard Treatment
Drug: Lip sunscreen 30 Sun Protector Factor (SPF) — Apply sunscreen on the lip 30 minutes every day before sun exposure. Protects against both UVA (ultraviolet A) and UVB (ultraviolet B rays).
Drug: Dexpanthenol — Apply dexpanthenol on the lip, two (2) times a day, once in the morning and once in the afternoon.
  Reduces transepidermic water loss and maintaining the natural smoothness and elasticity of the skin. It accelerates the cell renewal, rebuilds damaged tissues and promote the normal keratinisation of the skin and hair.

SUMMARY:
Actinic cheilitis is a potentially malignant lesion on the lower lip, which can progress to more serious illnesses such as cancer if not treated. Usually treatment of this condition is only based on clinical appearance, but there is no established cure treatment. Topical imiquimod is a medicine indicated for the treatment of skin diseases, but it has not yet been proven to treat actinic cheilitis. In this research, the investigator's aim is to evaluate the response to actinic cheilitis treatment with the current standard treatment compared to high and low concentration imiquimod topical formulations.

DETAILED DESCRIPTION:
Three formulations are used in this research: imiquimod 5%, imiquimod 0.05% e imiquimod nanoencapsulated 0.05%. Nanoencapsulation is a process that concentrates the drug into a capsule not visible to the naked eye, allowing it to penetrate skin more easily and will only release the drug at the lesion site. The drug is presented in a free form inside the gel in the others formulations.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with clinical and histopathological diagnosis of actinic cheilitis;
* No previous lip treatment with Imiquimod.

Exclusion Criteria:

* Present lesions suspected of squamous cell carcinoma of the lip.
* Previous history of lip cancer treatment.
* Prior treatment other than standard treatment.
* History of allergic reactions to imiquimod or any other component of the formulas.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Clinical Response | 30 days after conclusion of treatment
  Clinical analysis of lip photographs based on a classification. The lesions will be graded as:
  AC Grade I. Dryness and desquamation on the vermilion of lips.
  AC Grade II. Atrophy on the vermilion's border, presenting soft surfaces and pallid areas with eruptions. Blurred limit between the lip's vermilion border and the skin, or a dark line demarking that limit can be seen. This melanotic line should be different from ephelides or other pigmented lesions.
  AC Grade III. Rough and squamous areas on the drier parts of the vermilion and hyperkeratotic areas, especially when they spread to the wet lip's mucosa (border between mucosa and semimucosa).
  AC Grade IV. Ulceration present in one or more sites of the lip's vermillion or Leukoplakia, mainly in more traumatic places, due to the history of pipe or cigarettes consumption. These lesions could suggest that a malignization process would be in progress, especially when they are accompanied by endured areas on palpation.
Clinical Response | 180 days after conclusion of treatment
  Clinical analysis of lip photographs based on a classification. The lesions will be graded as:
  AC Grade I. Dryness and desquamation on the vermilion of lips.
  AC Grade II. Atrophy on the vermilion's border, presenting soft surfaces and pallid areas with eruptions. Blurred limit between the lip's vermilion border and the skin, or a dark line demarking that limit can be seen. This melanotic line should be different from ephelides or other pigmented lesions.
  AC Grade III. Rough and squamous areas on the drier parts of the vermilion and hyperkeratotic areas, especially when they spread to the wet lip's mucosa (border between mucosa and semimucosa).
  AC Grade IV. Ulceration present in one or more sites of the lip's vermillion or Leukoplakia, mainly in more traumatic places, due to the history of pipe or cigarettes consumption. These lesions could suggest that a malignization process would be in progress, especially when they are accompanied by endured areas on palpation.

SECONDARY OUTCOMES:
General Satisfaction about the medication: Visual Analogue Scale (VAS) | VAS scale will be generated at 14 days after beginning of the treatment.
  Satisfaction will be self-reported by VAS scale. The visual analogue scale (VAS) will be used to measure general satisfaction of participants to treatment. Participants will be asked to point in to a white paper with a 10cm line, where 0 represents none satisfaction and 10 maximum satisfaction.
General Satisfaction about the medication: Visual Analogue Scale (VAS) | VAS scale will be generated at 28 days after beginning of the treatment.
  Satisfaction will be self-reported by VAS scale. The visual analogue scale (VAS) will be used to measure general satisfaction of participants to treatment. Participants will be asked to point in to a white paper with a 10cm line, where 0 represents none satisfaction and 10 maximum satisfaction.
General Satisfaction about the medication: Visual Analogue Scale (VAS) | VAS scale will be generated at 60 days after beginning of the treatment.
  Satisfaction will be self-reported by VAS scale. The visual analogue scale (VAS) will be used to measure general satisfaction of participants to treatment. Participants will be asked to point in to a white paper with a 10cm line, where 0 represents none satisfaction and 10 maximum satisfaction.
General Satisfaction about the medication: Visual Analogue Scale (VAS) | VAS scale will be generated at 210 days after beginning of the treatment.
  Satisfaction will be self-reported by VAS scale. The visual analogue scale (VAS) will be used to measure general satisfaction of participants to treatment. Participants will be asked to point in to a white paper with a 10cm line, where 0 represents none satisfaction and 10 maximum satisfaction.
Adverse Events Severity | The adverse events questionnaire is applied in 14 days after beginning of the treatment.
  Adverse effects will be assessed during clinical evaluation at follow-up and with an adverse effects questionnaire.The questionnaire is based on self-reported events followed by a quantification of severity of local and systemic events. The participants are asked to classify the events in a scale of 0 to 3. 0= no sympton, 1- mild, 2-moderate and 3-severe.
Adverse Events Severity | The adverse events questionnaire is applied in 28 days after beginning of the treatment.
  Adverse effects will be assessed during clinical evaluation at follow-up and with an adverse effects questionnaire.The questionnaire is based on self-reported events followed by a quantification of severity of local and systemic events. The participants are asked to classify the events in a scale of 0 to 3. 0= no sympton, 1- mild, 2-moderate and 3-severe.
Adverse Events Severity | The adverse events questionnaire is applied in 60 days after beginning of the treatment.
  Adverse effects will be assessed during clinical evaluation at follow-up and with an adverse effects questionnaire.The questionnaire is based on self-reported events followed by a quantification of severity of local and systemic events. The participants are asked to classify the events in a scale of 0 to 3. 0= no sympton, 1- mild, 2-moderate and 3-severe.
Adverse Events Severity | The adverse events questionnaire is applied in 210 days after beginning of the treatment.
  Adverse effects will be assessed during clinical evaluation at follow-up and with an adverse effects questionnaire.The questionnaire is based on self-reported events followed by a quantification of severity of local and systemic events. The participants are asked to classify the events in a scale of 0 to 3. 0= no sympton, 1- mild, 2-moderate and 3-severe.
Maturation epithelial pattern | Maturation epithelial pattern analysis will be performed at 28 days after beginning of the treatment.
  Upon confirmation of the diagnosis of actinic cheilitis, participants will undergo a noninvasive procedure called exfoliative cytology. With this examination it is possible to analyze morphological changes of the collected cells by light microscopy. The lip mucosa is scraped with cytobrush, which is then used to smear two glass slides. From one of the obtained smears, Papanicolaou stain will be performed. Papanicoloau staining allows assessing different cell types, which are quantified to evaluate epithelial differentiation.
Maturation epithelial pattern | Maturation epithelial pattern analysis will be performed at 60 days after beginning of the treatment.
  Upon confirmation of the diagnosis of actinic cheilitis, participants will undergo a noninvasive procedure called exfoliative cytology. With this examination it is possible to analyze morphological changes of the collected cells by light microscopy. The lip mucosa is scraped with cytobrush, which is then used to smear two glass slides. From one of the obtained smears, Papanicolaou stain will be performed. Papanicoloau staining allows assessing different cell types, which are quantified to evaluate epithelial differentiation.
Maturation epithelial pattern | Maturation epithelial pattern analysis will be performed at 210 days after beginning of the treatment.
  Upon confirmation of the diagnosis of actinic cheilitis, participants will undergo a noninvasive procedure called exfoliative cytology. With this examination it is possible to analyze morphological changes of the collected cells by light microscopy. The lip mucosa is scraped with cytobrush, which is then used to smear two glass slides. From one of the obtained smears, Papanicolaou stain will be performed. Papanicoloau staining allows assessing different cell types, which are quantified to evaluate epithelial differentiation.
Cell proliferation - mAgNOR | mAgNOR analysis will be performed at 28 days after beginning of the treatment.
  Upon confirmation of the diagnosis of actinic cheilitis, participants will undergo a noninvasive procedure called exfoliative cytology. The lip mucosa is scraped with cytobrush, which is then used to smear two glass slides. One slide will be stained with AgNOR. With this examination it is possible to analyze cell proliferation activity. From the quantification of AgNORs, the average AgNORs / core (mAgNOR) will be calculated. The low average of AgNOR stained cells indicates lower cell proliferation and a higher average indicates greater proliferation.
Cell proliferation - mAgNOR | mAgNOR analysis will be performed at 60 days after beginning of the treatment.
  Upon confirmation of the diagnosis of actinic cheilitis, participants will undergo a noninvasive procedure called exfoliative cytology. The lip mucosa is scraped with cytobrush, which is then used to smear two glass slides. One slide will be stained with AgNOR. With this examination it is possible to analyze cell proliferation activity. From the quantification of AgNORs, the average AgNORs / core (mAgNOR) will be calculated. The low average of AgNOR stained cells indicates lower cell proliferation and a higher average indicates greater proliferation.
Cell proliferation - mAgNOR | mAgNOR analysis will be performed at 210 days after beginning of the treatment.
  Upon confirmation of the diagnosis of actinic cheilitis, participants will undergo a noninvasive procedure called exfoliative cytology. The lip mucosa is scraped with cytobrush, which is then used to smear two glass slides. One slide will be stained with AgNOR. With this examination it is possible to analyze cell proliferation activity. From the quantification of AgNORs, the average AgNORs / core (mAgNOR) will be calculated. The low average of AgNOR stained cells indicates lower cell proliferation and a higher average indicates greater proliferation.
Cell proliferation - pAgNOR | pAgNOR analysis will be performed at 28 days after beginning of the treatment.
  Upon confirmation of the diagnosis of actinic cheilitis, participants will undergo a noninvasive procedure called exfoliative cytology. The lip mucosa is scraped with cytobrush, which is then used to smear two glass slides. One slide will be stained with AgNOR. With this examination it is possible to analyze cell proliferation activity. A second evaluation parameter will be the percentage of cells with more than 1, 2, 3 and 4 AgNORs / nucleus (pAgNOR). A higher percentage of cells with more than 3 and 4 AgNORs per nucleus indicate greater proliferation.
Cell proliferation - pAgNOR | pAgNOR analysis will be performed at 60 days after beginning of the treatment.
  Upon confirmation of the diagnosis of actinic cheilitis, participants will undergo a noninvasive procedure called exfoliative cytology. The lip mucosa is scraped with cytobrush, which is then used to smear two glass slides. One slide will be stained with AgNOR. With this examination it is possible to analyze cell proliferation activity. A second evaluation parameter will be the percentage of cells with more than 1, 2, 3 and 4 AgNORs / nucleus (pAgNOR). A higher percentage of cells with more than 3 and 4 AgNORs per nucleus indicate greater proliferation.
Cell proliferation - pAgNOR | pAgNOR analysis will be performed at 210 days after beginning of the treatment.
  Upon confirmation of the diagnosis of actinic cheilitis, participants will undergo a noninvasive procedure called exfoliative cytology. The lip mucosa is scraped with cytobrush, which is then used to smear two glass slides. One slide will be stained with AgNOR. With this examination it is possible to analyze cell proliferation activity. A second evaluation parameter will be the percentage of cells with more than 1, 2, 3 and 4 AgNORs / nucleus (pAgNOR). A higher percentage of cells with more than 3 and 4 AgNORs per nucleus indicate greater proliferation.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Visioli, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (2):
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - School of Dentistry - Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poitevin NA, Rodrigues MS, Weigert KL, Macedo CLR, Dos Santos RB. Actinic cheilitis: proposition and reproducibility of a clinical criterion. BDJ Open. 2017 Aug 4;3:17016. doi: 10.1038/bdjopen.2017.16. eCollection 2017. PMID 29607086
- [Background] Bernardi A, Frozza RL, Jager E, Figueiro F, Bavaresco L, Salbego C, Pohlmann AR, Guterres SS, Battastini AM. Selective cytotoxicity of indomethacin and indomethacin ethyl ester-loaded nanocapsules against glioma cell lines: an in vitro study. Eur J Pharmacol. 2008 May 31;586(1-3):24-34. doi: 10.1016/j.ejphar.2008.02.026. Epub 2008 Feb 19. PMID 18371953
- [Background] Bernardi A, Zilberstein AC, Jager E, Campos MM, Morrone FB, Calixto JB, Pohlmann AR, Guterres SS, Battastini AM. Effects of indomethacin-loaded nanocapsules in experimental models of inflammation in rats. Br J Pharmacol. 2009 Oct;158(4):1104-11. doi: 10.1111/j.1476-5381.2009.00244.x. Epub 2009 May 6. PMID 19422380
- [Background] Bernardi A, Braganhol E, Jager E, Figueiro F, Edelweiss MI, Pohlmann AR, Guterres SS, Battastini AM. Indomethacin-loaded nanocapsules treatment reduces in vivo glioblastoma growth in a rat glioma model. Cancer Lett. 2009 Aug 18;281(1):53-63. doi: 10.1016/j.canlet.2009.02.018. Epub 2009 Mar 14. PMID 19286307
- [Background] Swanson N, Abramovits W, Berman B, Kulp J, Rigel DS, Levy S. Imiquimod 2.5% and 3.75% for the treatment of actinic keratoses: results of two placebo-controlled studies of daily application to the face and balding scalp for two 2-week cycles. J Am Acad Dermatol. 2010 Apr;62(4):582-90. doi: 10.1016/j.jaad.2009.07.004. Epub 2010 Feb 4. PMID 20133013
- [Background] Sotiriou E, Lallas A, Goussi C, Apalla Z, Trigoni A, Chovarda E, Ioannides D. Sequential use of photodynamic therapy and imiquimod 5% cream for the treatment of actinic cheilitis: a 12-month follow-up study. Br J Dermatol. 2011 Oct;165(4):888-92. doi: 10.1111/j.1365-2133.2011.10478.x. Epub 2011 Sep 15. PMID 21916880
- [Background] Smith KJ, Germain M, Yeager J, Skelton H. Topical 5% imiquimod for the therapy of actinic cheilitis. J Am Acad Dermatol. 2002 Oct;47(4):497-501. doi: 10.1067/mjd.2002.126266. PMID 12271290
- [Background] McDonald C, Laverick S, Fleming CJ, White SJ. Treatment of actinic cheilitis with imiquimod 5% and a retractor on the lower lip: clinical and histological outcomes in 5 patients. Br J Oral Maxillofac Surg. 2010 Sep;48(6):473-6. doi: 10.1016/j.bjoms.2009.08.024. PMID 19836865
- [Background] Manganaro AM, Will MJ, Poulos E. Actinic cheilitis: a premalignant condition. Gen Dent. 1997 Sep-Oct;45(5):492-4. PMID 9515418
- [Background] Lundeen RC, Langlais RP, Terezhalmy GT. Sunscreen protection for lip mucosa: a review and update. J Am Dent Assoc. 1985 Oct;111(4):617-21. doi: 10.14219/jada.archive.1985.0157. PMID 3877087
- [Background] Lebwohl M, Dinehart S, Whiting D, Lee PK, Tawfik N, Jorizzo J, Lee JH, Fox TL. Imiquimod 5% cream for the treatment of actinic keratosis: results from two phase III, randomized, double-blind, parallel group, vehicle-controlled trials. J Am Acad Dermatol. 2004 May;50(5):714-21. doi: 10.1016/j.jaad.2003.12.010. PMID 15097955
- [Background] Krawtchenko N, Roewert-Huber J, Ulrich M, Mann I, Sterry W, Stockfleth E. A randomised study of topical 5% imiquimod vs. topical 5-fluorouracil vs. cryosurgery in immunocompetent patients with actinic keratoses: a comparison of clinical and histological outcomes including 1-year follow-up. Br J Dermatol. 2007 Dec;157 Suppl 2:34-40. doi: 10.1111/j.1365-2133.2007.08271.x. PMID 18067630
- [Background] Kopera D, Kerl H. Visualization and treatment of subclinical actinic keratoses with topical imiquimod 5% cream: an observational study. Biomed Res Int. 2014;2014:135916. doi: 10.1155/2014/135916. Epub 2014 May 11. PMID 24900953
- [Background] Kaugars GE, Pillion T, Svirsky JA, Page DG, Burns JC, Abbey LM. Actinic cheilitis: a review of 152 cases. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1999 Aug;88(2):181-6. doi: 10.1016/s1079-2104(99)70115-0. PMID 10468463
- [Background] Jorizzo J, Dinehart S, Matheson R, Moore JK, Ling M, Fox TL, McRae S, Fielder S, Lee JH. Vehicle-controlled, double-blind, randomized study of imiquimod 5% cream applied 3 days per week in one or two courses of treatment for actinic keratoses on the head. J Am Acad Dermatol. 2007 Aug;57(2):265-8. doi: 10.1016/j.jaad.2007.01.047. Epub 2007 May 18. PMID 17512087
- [Background] Greenberg HL, Cohen JL, Rosen T, Orengo I. Severe reaction to 5% imiquimod cream with excellent clinical and cosmetic outcomes. J Drugs Dermatol. 2007 Apr;6(4):452-8. PMID 17668546
- [Background] Gebauer K, Shumack S, Cowen PS. Effect of dosing frequency on the safety and efficacy of imiquimod 5% cream for treatment of actinic keratosis on the forearms and hands: a phase II, randomized placebo-controlled trial. Br J Dermatol. 2009 Oct;161(4):897-903. doi: 10.1111/j.1365-2133.2009.09260.x. Epub 2009 May 26. PMID 19545297
- [Background] A Gaspari A, Tyring SK, Rosen T. Beyond a decade of 5% imiquimod topical therapy. J Drugs Dermatol. 2009 May;8(5):467-74. PMID 19537370
- [Background] Frank LA, Chaves PS, D'Amore CM, Contri RV, Frank AG, Beck RC, Pohlmann AR, Buffon A, Guterres SS. The use of chitosan as cationic coating or gel vehicle for polymeric nanocapsules: Increasing penetration and adhesion of imiquimod in vaginal tissue. Eur J Pharm Biopharm. 2017 May;114:202-212. doi: 10.1016/j.ejpb.2017.01.021. Epub 2017 Feb 1. PMID 28161547
- [Background] Frank LA, Sandri G, D'Autilia F, Contri RV, Bonferoni MC, Caramella C, Frank AG, Pohlmann AR, Guterres SS. Chitosan gel containing polymeric nanocapsules: a new formulation for vaginal drug delivery. Int J Nanomedicine. 2014 Jun 28;9:3151-61. doi: 10.2147/IJN.S62599. eCollection 2014. PMID 25061292
- [Background] Ferreira AM, de Souza Lucena EE, de Oliveira TC, da Silveira E, de Oliveira PT, de Lima KC. Prevalence and factors associated with oral potentially malignant disorders in Brazil's rural workers. Oral Dis. 2016 Sep;22(6):536-42. doi: 10.1111/odi.12488. Epub 2016 May 17. PMID 27090966
- [Background] Falagas ME, Angelousi AG, Peppas G. Imiquimod for the treatment of actinic keratosis: A meta-analysis of randomized controlled trials. J Am Acad Dermatol. 2006 Sep;55(3):537-8. doi: 10.1016/j.jaad.2006.05.030. No abstract available. PMID 16908371
- [Background] Eigentler TK, Kamin A, Weide BM, Breuninger H, Caroli UM, Mohrle M, Radny P, Garbe C. A phase III, randomized, open label study to evaluate the safety and efficacy of imiquimod 5% cream applied thrice weekly for 8 and 12 weeks in the treatment of low-risk nodular basal cell carcinoma. J Am Acad Dermatol. 2007 Oct;57(4):616-21. doi: 10.1016/j.jaad.2007.05.022. Epub 2007 Jul 3. PMID 17610993
- [Background] Dufresne RG Jr, Curlin MU. Actinic cheilitis. A treatment review. Dermatol Surg. 1997 Jan;23(1):15-21. PMID 9107289
- [Background] dos Santos LR, Cernea CR, Kowalski LP, Carneiro PC, Soto MN, Nishio S, Hojaij FC, Dutra Junior A, Britto e Silva Filho G, Ferraz AR. Squamous-cell carcinoma of the lower lip: a retrospective study of 58 patients. Sao Paulo Med J. 1996 Mar-Apr;114(2):1117-26. doi: 10.1590/s1516-31801996000200003. PMID 9077021
- [Background] Daniel FI, Alves SR, Vieira DS, Biz MT, Daniel IW, Modolo F. Immunohistochemical expression of DNA methyltransferases 1, 3a, and 3b in actinic cheilitis and lip squamous cell carcinomas. J Oral Pathol Med. 2016 Nov;45(10):774-779. doi: 10.1111/jop.12453. Epub 2016 May 9. PMID 27159259
- [Background] de Souza Lucena EE, Costa DC, da Silveira EJ, Lima KC. Prevalence and factors associated to actinic cheilitis in beach workers. Oral Dis. 2012 Sep;18(6):575-9. doi: 10.1111/j.1601-0825.2012.01910.x. Epub 2012 Feb 15. PMID 22335283
- [Background] Contri RV, Katzer T, Ourique AF, da Silva AL, Beck RC, Pohlmann AR, Guterres SS. Combined effect of polymeric nanocapsules and chitosan hydrogel on the increase of capsaicinoids adhesion to the skin surface. J Biomed Nanotechnol. 2014 May;10(5):820-30. doi: 10.1166/jbn.2014.1752. PMID 24734535
- [Background] Couvreur P, Barratt G, Fattal E, Legrand P, Vauthier C. Nanocapsule technology: a review. Crit Rev Ther Drug Carrier Syst. 2002;19(2):99-134. doi: 10.1615/critrevtherdrugcarriersyst.v19.i2.10. PMID 12197610
- [Background] Contri RV, Frank LA, Kaiser M, Pohlmann AR, Guterres SS. The use of nanoencapsulation to decrease human skin irritation caused by capsaicinoids. Int J Nanomedicine. 2014 Feb 12;9:951-62. doi: 10.2147/IJN.S56579. eCollection 2014. PMID 24611011
- [Background] Cavalcante AS, Anbinder AL, Carvalho YR. Actinic cheilitis: clinical and histological features. J Oral Maxillofac Surg. 2008 Mar;66(3):498-503. doi: 10.1016/j.joms.2006.09.016. PMID 18280383
- [Background] Cataldo E, Doku HC. Solar cheilitis. J Dermatol Surg Oncol. 1981 Dec;7(12):989-95. doi: 10.1111/j.1524-4725.1981.tb00203.x. PMID 7338591
- [Background] Bulcao RP, Freitas FA, Venturini CG, Dallegrave E, Durgante J, Goethel G, Cerski CT, Zielinsky P, Pohlmann AR, Guterres SS, Garcia SC. Acute and subchronic toxicity evaluation of poly(epsilon-caprolactone) lipid-core nanocapsules in rats. Toxicol Sci. 2013 Mar;132(1):162-76. doi: 10.1093/toxsci/kfs334. Epub 2012 Dec 12. PMID 23235194
- [Background] Bulcao RP, de Freitas FA, Dallegrave E, Venturini CG, Baierle M, Durgante J, Sauer E, Cassini C, Cerski CT, Zielinsky P, Salvador M, Pohlmann AR, Guterres SS, Garcia SC. In vivo toxicological evaluation of polymeric nanocapsules after intradermal administration. Eur J Pharm Biopharm. 2014 Feb;86(2):167-77. doi: 10.1016/j.ejpb.2013.04.001. Epub 2013 May 2. PMID 23643792
- [Background] Spyridonos P, Gaitanis G, Tzaphlidou M, Bassukas ID. Spatial fuzzy c-means algorithm with adaptive fuzzy exponent selection for robust vermilion border detection in healthy and diseased lower lips. Comput Methods Programs Biomed. 2014 May;114(3):291-301. doi: 10.1016/j.cmpb.2014.02.017. Epub 2014 Mar 6. PMID 24661607
- [Derived] da Silva EL, Pedraca ES, Salgueiro AP, Gazzi RP, Nunes JS, Cavagni J, Martins MAT, Rados PV, Pohlmann AR, Guterres SS, Frank LA, Visioli F. Efficacy and safety of a 0.05 % nanoencapsulated imiquimod hydrogel for the treatment of actinic cheilitis: Drug release analysis and clinical study. Nanomedicine. 2024 Nov;62:102779. doi: 10.1016/j.nano.2024.102779. Epub 2024 Aug 14. PMID 39147219